CLINICAL TRIAL: NCT05251922
Title: Tolerance of Anti-Cancer Therapy in the Elderly
Acronym: TOASTIE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: MO19/127559
Record Dates: First submitted 2022-01-26; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Frailty; Chemotherapeutic Toxicity
Keywords: frailty; chemotherapy tolerance
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicentre observational study evaluating frailty and tolerance of chemotherapy in the elderly.

DETAILED DESCRIPTION:
This is a multicentre observational study evaluating frailty and tolerance of chemotherapy in the elderly.

The number of people with cancer over the age of 65 years is increasing and more older patients are being treated with chemotherapy. Previous research has shown that patients living with frailty are more likely to experience significant toxicity from chemotherapy.

A scoring system exists, the CARG (Cancer Aging Research Group) score), which using sociodemographics, tumour/treatment variables, laboratory test results (haemoglobin and creatinine clearance), geriatric assessment variables (function, co-morbidity, cognition, psychological state, social activity/support and nutritional status) predicts the likelihood of patients in this population developing a grade 3-5 toxicity. The CARG score ranges from 0 (lowest toxicity risk) to 19 (highest toxicity risk).

This scoring system was developed and validated in the USA (United States of America). It was not however found to be predictive of toxicity in Australia. To date it has not been evaluated, nor is used in routine practice in oncology in the UK (United Kingdom).

This study is looking at markers of frailty in patients >65years. The investigators seek to predict those who are at a higher risk of side effects from chemotherapy. The investigators are looking to validate the CARG score in a UK NHS (National Health Service) population and show feasibility of using this in routine practice. The investigators are also evaluating if other scoring systems which are routinely used to assess frailty (but have never been assessed for predicting toxicity) are useful in predicting toxicity.

Secondary objectives include describing frailty in this population, exploring patients' perceptions of risk associated with chemotherapy and demonstrating the added value of risk prediction tools compared to clinicians estimates of toxicity risk.

ELIGIBILITY:
Inclusion Criteria:

* Age >65years
* About to start first line chemotherapy for a solid tumour based malignancy
* Chemotherapy given for any intent eg. adjuvant or palliative
* Estimated survival of >3months
* Able to comprehend and complete questionnaire.

Exclusion Criteria:

* Medical or psychiatric condition impairing ability to consent
* Participant is enrolled in another clinical trial
* Prior chemotherapy for any indication
* Receiving concurrent radiotherapy (RT) or immunotherapy (IT)
* Unable to provide informed consent

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Adults aged 65years or over, about to receive first line chemotherapy for a solid tumour based malignancy
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
To validate the CARG scoring system | 6 months follow up
  To validate the CARG scoring system (a score which is calculated by the doctor using patient information) in a UK real-world population and show feasibility of implementing CARG scoring in routine NHS practice.
  The investigators will collect the information required and calculate a CARG score for each participant.
  The investigators will record Grade 3-5 chemotherapy toxicities (as assessed using CTCAEv5) for each participant.
  The investigators will evaluate if the CARG score is predictive of Grade 3-5 toxicity (as assessed using CTCAEv5) in this UK real-world population.
  The investigators will record how long it takes to collect this information and calculate the score to see if it is feasible to implement this in a real world setting.

SECONDARY OUTCOMES:
Describe frailty in elderly patients (>65years) in the UK NHS prior to starting chemotherapy - demographics | 6 months follow up
  The investigators are reporting demographics: age (years) and gender
Describe frailty in elderly patients (>65years) in the UK NHS prior to starting chemotherapy - tumour type | 6 months follow up
  The investigators are reporting tumour type eg. breast cancer, gastric cancer etc.
Describe frailty in elderly patients (>65years) in the UK NHS prior to starting chemotherapy - chemotherapy type | 6 months follow up
  The investigators will be reporting chemotherapy drugs delivered
Describe frailty in elderly patients (>65years) in the UK NHS prior to starting chemotherapy - laboratory test results (Hb) | 6 months follow up
  The investigators will be reporting laboratory test results prior to first cycle of chemotherapy
  -haemoglobin (g/L)
Describe frailty in elderly patients (>65years) in the UK NHS prior to starting chemotherapy - laboratory test results (CrCl) | 6 months follow up
  The investigators will be reporting laboratory test results prior to first cycle of chemotherapy
  -creatinine clearance (mL/min)
Describe frailty in elderly patients (>65years) in the UK NHS prior to starting chemotherapy using SIOG (International Society of Geriatric Oncology) Geriatric Screening Tool (G8) | 6 months follow up
  Investigators will calculate the SIOG (International Society of Geriatric Oncology) Geriatric Screening Tool (G8) and report the score
Describe frailty in elderly patients (>65years) in the UK NHS prior to starting chemotherapy using the Rockwood Clinical Frailty Score (CFS) | 6 months follow up
  Investigators will record the Rockwood Clinical Frailty Score (CFS) and report the scores
Evaluate the predictive value of commonly used geriatric assessment tools in predicting chemotherapy tolerance | 6 months follow up
  Frailty scoring systems (G8 and CFS) will be calculated. Grade 3-5 chemotherapy toxicities will (as assessed using CTCAEv5) will be recorded.
  The investigators will assess if these scoring systems have utility in predicting risk of grade 3-5 chemotherapy toxicity.
The CARG score which reports the risk of grade 3-5 toxicity as assessed using CTCAEv5 as a percentage. | 6 months follow up
Explore patients perception of risk associated with chemotherapy in this population | 6 months follow up
  Participants will report their perception of likelihood of developing a side effect from chemotherapy which would cause the participant to stay in hospital for one night or longer or have to stop treatment using the following options: Unlikely, Not very likely, Quite likely or Very likely, as well as using a percentage scale as seen below.
  0 means I think it definitely won't happen to me → 100 means I think I will definitely need to stop treatment or stay hospital at some point during my treatment
  0-----10-----20-----30-----40-----50-----60-----70-----80-----90----100

CONTACTS AND LOCATIONS:
Overall Officials: Helen C Dearden, Principal Investigator — helen.dearden1@nhs.net
Locations (1):
- Leeds NHS Teaching Hospitals, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No